CLINICAL TRIAL: NCT06131619
Title: The Role of Dynamic Lowenstein Occupational Therapy Cognitive Assessment-Geriatric Version (DLOTCA-G) in the Cognitive Function Evaluation of Parkinson's Patients
Brief Title: The Role of DLOTCA-G in the Cognitive Function Evaluation of Parkinson's Patients
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Merve Akdeniz Leblebicier, assoc.prof dr, Kutahya Health Sciences University
Other Study IDs: 2021/15-03
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; DLOTCA-G
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental: Parkinson's disease patients with cognitive impairment
  Interventions: Other: assesment of cognitive parameters with DLOTCA-G
- Active Comparator: Parkinson's disease patients without cognıtıve impairment
  Interventions: Other: assesment of cognitive parameters with DLOTCA-G
- other: Health geriatric persons
  Interventions: Other: assesment of cognitive parameters with DLOTCA-G

INTERVENTIONS:
Other: assesment of cognitive parameters with DLOTCA-G — All three groups were evaluated once with the DLOTCA-G, a cognitive assessment battery.

SUMMARY:
The purpose of this study is to evaluate the usefulness of Dynamic Loewenstein's Occupational Therapy and Cognitive Assessment Scale for Geriatrics (DLOTCA-G) in parkinson patients.

DETAILED DESCRIPTION:
The purpose of this study to evaluate the usefulness of Dynamic Loewenstein's Occupational Therapy and Cognitive Assessment Scale for Geriatrics (DLOTCA-G) in the early detection of cognitive impairment in parkinson patients aged 65 and over, with and without dementia.The investigators also aimed to compare the Mini Mental State Assessment Test with DLOTCA-G.

ELIGIBILITY:
Inclusıon Criteria

* Parkinson's patients aged 65 years and older with and without cognitive impairment (60 patients) and healthy control patients (30 patients)
* Hoehnn Yahr Staging between 1 and 2.5 in patients with Parkinson's diseas
* Confirmed by brain MRI from patients without vascular dementia who routinely attend the Parkinson's follow-up outpatient clinic
* At least primary school graduates
* In patients with Parkinson's dissease patients with cognitive impairment, MMSE below 20 in primary school education level; below 24 in secondary, high school and university education level
* In patients with Parkinson's disease without cognitive impairment, MMSE 20 and above in primary school education level; 24 and above in secondary, high school and university education level Exclusıon Criteria
* Preexisting cognitive impairment
* Psychiatric disorders such as psychotic disorders, mood disorders, alcohol or drug abuse
* Severe language dysfunction and/or bilateral limb motor dysfunction and inability to participate in clinical psychology tests, severe visual and/or auditory impairments
* Patients with significant cerebral atrophy or neurological vascular lesions
* The Geriatric Depression Scale was administered to all participants, and participants with a total score of 13 or more out of 30 points were excluded from the study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Parkinson's dissease patients
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Dynamic Lowenstein Occupational Therapy Cognitive Assessment-Geriatric Version | Baseline (First assessment)
  The Dynamic Lowenstein Occupational Therapy Cognitive Assessment is an occupational performance measurement battery designed to assess basic cognitive skills and visual perception in adults with neurological deficits. Consists 8 subtests: orientation, awareness, visual perception, spatial perception, praxis, visuomotor construction and thinking operations and memory. All subtests of DLOTCA-G are scored between 1 - 4 points. And higher scores indicate better cognitive performance. There is no cut-off value for Parkinson's patients.

SECONDARY OUTCOMES:
Mini Mental State Examination | Baseline (First assessment)
  The Mini Mental State Examination is a brief screening tool that provides a quantitative assessment of cognitive impairment and to record cognitive changes over time. It consists of five subscales: orientation, memory, attention and calculation, recall and language. In the evaluation of the test, scores below 15 indicate low cognitive level, scores between 15 and 26 indicate medium cognitive level, and scores of 26 and above indicate high cognitive level.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)